CLINICAL TRIAL: NCT05185622
Title: A Phase II Open-Label, Multiple Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Exploratory Efficacy of Vamorolone in Boys Ages 2 to <4 Years and 7 to <18 Years With Duchenne Muscular Dystrophy (DMD)
Brief Title: A Study to Assess Vamorolone in Boys Ages 2 to <4 Years and 7 to <18 Years With Duchenne Muscular Dystrophy (DMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VBP15-006
Expanded Access: NCT03863119 (Available)
Record Dates: First submitted 2021-11-09; First posted 2022-01-11 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-09

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy; Duchenne and Becker Muscular Dystrophy; Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies | interventions — VBP15 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Treatment Group 1 (Experimental): Patients in Treatment Group 1 must be ages 2-<4 years and will receive Vamorolone at 2.0 mg/kg/day for the duration of the study. Treatment Group 1 will be enrolled prior to Treatment Group 2.
  Interventions: Drug: Vamorolone
- Treatment Group 2 (Experimental): Patients in Treatment Group 2 must be ages 2-<4 years and will receive Vamorolone at 6.0 mg/kg/day for the duration of the study. Treatment Group 2 will be enrolled after Treatment Group 1.
  Interventions: Drug: Vamorolone
- Treatment Group 3 (Experimental): Patients in Treatment Group 3 must be ages 7-<18 years and must be steroid untreated at entry. Treatment Group 3 will receive Vamorolone at 2.0 mg/kg/day for the duration of the study.
  Interventions: Drug: Vamorolone
- Treatment Group 4 (Experimental): Patients in Treatment Group 4 must be ages 7-<18 years and must be steroid untreated at entry. Treatment Group 4 will receive Vamorolone at 6.0 mg/kg/day for the duration of the study.
  Interventions: Drug: Vamorolone
- Treatment Group 5 (Experimental): Patients in Treatment Group 5 must be ages 7-<18 years and must be on a stable dose of steroid for 3 months prior to entry. Treatment Group 5 will receive Vamorolone at 2.0 mg/kg/day for the duration of the study.
  Interventions: Drug: Vamorolone
- Treatment Group 6 (Experimental): Patients in Treatment Group 6 must be ages 7-<18 years and must be on a stable dose of steroid for 3 months prior to entry. Treatment Group 6 will receive Vamorolone at 6.0 mg/kg/day for the duration of the study.
  Interventions: Drug: Vamorolone
- Treatment Sub-Group 7 (Experimental): Patients in Treatment Sub-Group 7 must be ages 12-<18 years and must be on a stable dose of steroid for 3 months prior to entry. Treatment Group 7 will receive Vamorolone at 6.0 mg/kg/day for the duration of the study.
  Interventions: Drug: Vamorolone

INTERVENTIONS:
Drug: Vamorolone — Oral administration of vamorolone for 12 weeks.
  Other Names: VBP15

SUMMARY:
This Phase II study is an open-label, multiple dose study to evaluate the safety, tolerability, PK, PD, clinical efficacy, behavior and neuropsychology, and physical functioning vamorolone over a treatment period of 12 weeks in steroid-naïve boys ages 2 to <4 years, and glucocorticoid-treated and currently untreated boys ages 7 to <18 years with DMD.

DETAILED DESCRIPTION:
This Phase II study is an open-label, multiple dose study to evaluate the safety, tolerability, PK, PD, clinical efficacy, behavior and neuropsychology, and physical functioning of vamorolone administered orally at daily doses of 2.0 mg/kg and 6.0 mg/kg over a treatment period of 3 months in steroid-naïve boys ages 2 to <4, and glucocorticoid-treated and currently untreated boys ages 7 to <18 years with DMD.

The study is comprised of a 5-week Pretreatment Screening Period; a 1-day Pretreatment Baseline Period; a 3-month open-label Treatment Period (Weeks 1-12); and a 4-8 week open-label Dose-tapering Period (starting from Weeks 13) for subjects who will not transition directly to further vamorolone or standard of care (SoC) glucocorticoid treatment at the end of the study.

Subjects will be enrolled into the study at the Screening Visit, at the time written informed consent is obtained.

Within the 2 to <4 years age group, the initial 10 eligible subjects will be assigned to the 2.0 mg/kg/day treatment group at the Baseline Day -1 Visit. The subsequent 10 eligible subjects will be assigned to the 6.0 mg/kg/day treatment group at the Baseline Day -1 Visit.

Within the 7 to <18 years age group, both corticosteroid-treated and untreated, the initial 12 eligible subjects will be assigned to the 2.0 mg/kg/day treatment group at the Baseline Day -1 Visit. The subsequent 12 eligible subjects will be assigned to the 6.0 mg/kg/day treatment group at the Baseline Day -1 Visit.

The first 6 subjects in each age group at 2 mg/kg will serve as the PK/safety run-in cohorts. PK assessments will be performed at week 2 and together with the safety assessment during the first 4 weeks of treatment this will be the basis to confirm whether 2 and 6 mg/kg/day will be used in the subsequent patients or if a dose adjustment is needed to avoid over or under-exposure in patients for any of the two age groups.

Glucocorticoid-treated subjects in the 7 to <18 years age group will take their final dose of SoC glucocorticoid therapy for DMD on Baseline Day -1, within 24 hours prior to administration of the first dose of vamorolone study medication.

All subjects in both age groups will begin their assigned vamorolone treatment on Treatment Period Day 1, and will continue to receive their assigned vamorolone treatment throughout the duration of the 3 month Treatment Period (Weeks 1-12).

At the end of the 3-month Treatment Period (Week 12), subjects will be given the option to receive vamorolone in an expanded access or compassionate use program, if possible, or to transition to SoC treatment for DMD (may include glucocorticoids). Subjects completing VBP15-006 and enrolling directly into the expanded access or compassionate use program or transitioning directly to SoC glucocorticoid treatment will not need to taper their vamorolone dose prior to participation in the expanded access or compassionate use program or initiation of SoC glucocorticoid treatment. All subjects who will not transition directly to further vamorolone or SoC glucocorticoid treatment will begin a 4 -8 week open label Dose tapering Period during which the dose of study medication will be progressively reduced and discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's parent(s) or legal guardian(s) has (have) provided written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization, where applicable, prior to any study-related procedures; participants will be asked to give written or verbal assent according to local requirements;
2. Subject has a centrally confirmed (by TRiNDS central genetic counselor[s]) diagnosis of DMD, defined as:

   1. Dystrophin immunofluorescence and/or immunoblot showing complete dystrophin deficiency, and clinical picture consistent with typical DMD, OR
   2. Identifiable mutation within the DMD gene (deletion/duplication of one or more exons), where reading frame can be predicted as 'out-of-frame,' and clinical picture consistent with typical DMD, OR
   3. Complete dystrophin gene sequencing showing an alteration (point mutation, duplication, other) that is expected to preclude production of the dystrophin protein (i.e., nonsense mutation, deletion/duplication leading to a downstream stop codon), with a clinical picture consistent with typical DMD;
3. Subject is male, 2 to <4 years or 7 to <18 years of age at time of enrollment in the study;
4. If 7 to <18 years of age and currently taking standard of care glucocorticoids for treatment of DMD, subject has been taking standard of care glucocorticoids at stable dose for at least 3 months prior to enrollment in the study, and will continue the same stable dose regimen through the date of the Baseline Day -1 Visit. [Note: Inhaled and/or topical glucocorticoids are permitted if last use is at least 4 weeks prior to enrollment or if administered at stable dose beginning at least 4 weeks prior to enrollment and anticipated to be used at the stable dose regimen for the duration of the study];
5. If 7 to <18 years of age, and not currently glucocorticoid-treated, subject has not received oral glucocorticoids or other oral immunosuppressive agents for at least 3 months prior to enrollment. [Note: Inhaled and/or topical glucocorticoids are permitted if last use is at least 4 weeks prior to enrollment or if administered at stable dose beginning at least 4 weeks prior to enrollment and anticipated to be used at the stable dose regimen for the duration of the study];
6. Clinical laboratory test results are within the normal range at the Screening Visit, or if abnormal, are not clinically significant, in the opinion of the Investigator. [Notes: Serum gamma glutamyl transferase (GGT), creatinine, and total bilirubin all must be ≤ upper limit of the normal range at the Screening Visit. An abnormal vitamin D level that is considered clinically significant will not exclude a subject from participating];
7. Subject has evidence of chicken pox immunity as determined by:

   * Presence of IgG antibodies to varicella, as documented by a positive test result from the local laboratory from blood collected during the Screening Period; OR
   * Documentation, provided at the Screening Visit, that the subject has had 2 doses of varicella vaccine, with or without serologic evidence of immunity; the second of the 2 immunizations must have been given at least 14 days prior to assignment to a dose group;
8. Subject and parent(s)/guardian(s) are willing and able to comply with scheduled visits, study drug administration plan, and study procedures.

Exclusion Criteria:

1. Subject has current or history of major renal or hepatic impairment, diabetes mellitus or immunosuppression;
2. Subject has current or history of chronic systemic fungal or viral infections;
3. Subject has used mineralocorticoid receptor agents, such as spironolactone, eplerenone, canrenone (canrenoate potassium), prorenone (prorenoate potassium), or mexrenone (mexrenoate potassium) within 4 weeks prior to enrollment;
4. Subject has a history of primary hyperaldosteronism;
5. Subject has evidence of symptomatic cardiomyopathy [Note: Asymptomatic cardiac abnormality on investigation would not be exclusionary];
6. If 2 to <4 years of age, subject is currently being treated or has received previous treatment with oral glucocorticoids or other immunosuppressive agents [Notes: Past transient use of oral glucocorticoids or other oral immunosuppressive agents for no longer than 1 month cumulative, with last use at least 3 months prior to enrollment, will be considered for eligibility on a case-by-case basis, unless discontinued for intolerance. Inhaled and/or topical glucocorticoids are permitted if last use is at least 4 weeks prior to enrollment or if administered at stable dose beginning at least 4 weeks prior to enrollment and anticipated to be used at the stable dose regimen for the duration of the study];
7. Subject has an allergy or hypersensitivity to the study medication or to any of its constituents;
8. Subject has used idebenone within 4 weeks prior to enrollment;
9. Subject has severe behavioral or cognitive problems that preclude participation in the study, in the opinion of the Investigator;
10. Subject has previous or ongoing medical condition, medical history, physical findings or laboratory abnormalities that could affect safety, make it unlikely that treatment and follow-up will be correctly completed or impair the assessment of study results, in the opinion of the Investigator;
11. Subject is taking (or has taken within 4 weeks prior to enrollment) herbal remedies and supplements which can impact muscle strength and function (e.g., Co-enzyme Q10, creatine, etc);
12. Subject is taking (or has taken within 3 months prior to enrollment) any medication indicated for DMD, including Exondys51, Exondys53, Exondys45, Viltepso and Translarna;
13. Subject has been administered a live attenuated vaccine within 14 days prior to the first dose of study medication;
14. Subject is currently taking any other investigational drug or has taken any other investigational drug within 3 months prior to enrollment;
15. Subject has previously been enrolled in the VBP15-006 study or any other vamorolone study.

Ages: 2 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean K Mah, M.D., Principal Investigator — Alberta Children's Hospital Research Institute, University of Calgary
Locations (5):
- Canada (5):
  - Alberta's Children Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Montreal Childrens Hospital, Montreal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoffman EP, Schwartz BD, Mengle-Gaw LJ, Smith EC, Castro D, Mah JK, McDonald CM, Kuntz NL, Finkel RS, Guglieri M, Bushby K, Tulinius M, Nevo Y, Ryan MM, Webster R, Smith AL, Morgenroth LP, Arrieta A, Shimony M, Siener C, Jaros M, Shale P, McCall JM, Nagaraju K, van den Anker J, Conklin LS, Cnaan A, Gordish-Dressman H, Damsker JM, Clemens PR; Cooperative International Neuromuscular Research Group. Vamorolone trial in Duchenne muscular dystrophy shows dose-related improvement of muscle function. Neurology. 2019 Sep 24;93(13):e1312-e1323. doi: 10.1212/WNL.0000000000008168. Epub 2019 Aug 26. PMID 31451516
- [Background] Smith EC, Conklin LS, Hoffman EP, Clemens PR, Mah JK, Finkel RS, Guglieri M, Tulinius M, Nevo Y, Ryan MM, Webster R, Castro D, Kuntz NL, Kerchner L, Morgenroth LP, Arrieta A, Shimony M, Jaros M, Shale P, Gordish-Dressman H, Hagerty L, Dang UJ, Damsker JM, Schwartz BD, Mengle-Gaw LJ, McDonald CM; CINRG VBP15 and DNHS Investigators. Efficacy and safety of vamorolone in Duchenne muscular dystrophy: An 18-month interim analysis of a non-randomized open-label extension study. PLoS Med. 2020 Sep 21;17(9):e1003222. doi: 10.1371/journal.pmed.1003222. eCollection 2020 Sep. PMID 32956407
- [Background] Heier CR, Yu Q, Fiorillo AA, Tully CB, Tucker A, Mazala DA, Uaesoontrachoon K, Srinivassane S, Damsker JM, Hoffman EP, Nagaraju K, Spurney CF. Vamorolone targets dual nuclear receptors to treat inflammation and dystrophic cardiomyopathy. Life Sci Alliance. 2019 Feb 11;2(1):e201800186. doi: 10.26508/lsa.201800186. Print 2019 Feb. PMID 30745312
- [Background] Mavroudis PD, van den Anker J, Conklin LS, Damsker JM, Hoffman EP, Nagaraju K, Clemens PR, Jusko WJ. Population Pharmacokinetics of Vamorolone (VBP15) in Healthy Men and Boys With Duchenne Muscular Dystrophy. J Clin Pharmacol. 2019 Jul;59(7):979-988. doi: 10.1002/jcph.1388. Epub 2019 Feb 11. PMID 30742306
- [Background] Damsker JM, Cornish MR, Kanneboyina P, Kanneboyina I, Yu Q, Lipson R, Phadke A, Knoblach SM, Panchapakesan K, Morales M, Fiorillo AA, Partridge T, Nagaraju K. Vamorolone, a dissociative steroidal compound, reduces collagen antibody-induced joint damage and inflammation when administered after disease onset. Inflamm Res. 2019 Nov;68(11):969-980. doi: 10.1007/s00011-019-01279-z. Epub 2019 Aug 24. PMID 31446438
- [Background] Akkad H, Cacciani N, Llano-Diez M, Corpeno Kalamgi R, Tchkonia T, Kirkland JL, Larsson L. Vamorolone treatment improves skeletal muscle outcome in a critical illness myopathy rat model. Acta Physiol (Oxf). 2019 Feb;225(2):e13172. doi: 10.1111/apha.13172. Epub 2018 Sep 6. PMID 30120816
- [Background] Li X, Conklin LS, van den Anker J, Hoffman EP, Clemens PR, Jusko WJ. Exposure-Response Analysis of Vamorolone (VBP15) in Boys With Duchenne Muscular Dystrophy. J Clin Pharmacol. 2020 Oct;60(10):1385-1396. doi: 10.1002/jcph.1632. Epub 2020 May 20. PMID 32434278
- [Background] Hoffman EP, Riddle V, Siegler MA, Dickerson D, Backonja M, Kramer WG, Nagaraju K, Gordish-Dressman H, Damsker JM, McCall JM. Phase 1 trial of vamorolone, a first-in-class steroid, shows improvements in side effects via biomarkers bridged to clinical outcomes. Steroids. 2018 Jun;134:43-52. doi: 10.1016/j.steroids.2018.02.010. Epub 2018 Mar 8. PMID 29524454
- [Background] Almeida LEF, Damsker JM, Albani S, Afsar N, Kamimura S, Pratt D, Kleiner DE, Quezado M, Gordish-Dressman H, Quezado ZMN. The corticosteroid compounds prednisolone and vamorolone do not alter the nociception phenotype and exacerbate liver injury in sickle cell mice. Sci Rep. 2018 Apr 17;8(1):6081. doi: 10.1038/s41598-018-24274-6. PMID 29666400
- [Background] Wells E, Kambhampati M, Damsker JM, Gordish-Dressman H, Yadavilli S, Becher OJ, Gittens J, Stampar M, Packer RJ, Nazarian J. Vamorolone, a dissociative steroidal compound, reduces pro-inflammatory cytokine expression in glioma cells and increases activity and survival in a murine model of cortical tumor. Oncotarget. 2017 Feb 7;8(6):9366-9374. doi: 10.18632/oncotarget.14070. PMID 28030841
- [Background] Conklin LS, Damsker JM, Hoffman EP, Jusko WJ, Mavroudis PD, Schwartz BD, Mengle-Gaw LJ, Smith EC, Mah JK, Guglieri M, Nevo Y, Kuntz N, McDonald CM, Tulinius M, Ryan MM, Webster R, Castro D, Finkel RS, Smith AL, Morgenroth LP, Arrieta A, Shimony M, Jaros M, Shale P, McCall JM, Hathout Y, Nagaraju K, van den Anker J, Ward LM, Ahmet A, Cornish MR, Clemens PR. Phase IIa trial in Duchenne muscular dystrophy shows vamorolone is a first-in-class dissociative steroidal anti-inflammatory drug. Pharmacol Res. 2018 Oct;136:140-150. doi: 10.1016/j.phrs.2018.09.007. Epub 2018 Sep 13. PMID 30219580
- [Background] Fiorillo AA, Tully CB, Damsker JM, Nagaraju K, Hoffman EP, Heier CR. Muscle miRNAome shows suppression of chronic inflammatory miRNAs with both prednisone and vamorolone. Physiol Genomics. 2018 Sep 1;50(9):735-745. doi: 10.1152/physiolgenomics.00134.2017. Epub 2018 Jun 8. PMID 29883261
- [Background] Sreetama SC, Chandra G, Van der Meulen JH, Ahmad MM, Suzuki P, Bhuvanendran S, Nagaraju K, Hoffman EP, Jaiswal JK. Membrane Stabilization by Modified Steroid Offers a Potential Therapy for Muscular Dystrophy Due to Dysferlin Deficit. Mol Ther. 2018 Sep 5;26(9):2231-2242. doi: 10.1016/j.ymthe.2018.07.021. Epub 2018 Aug 27. PMID 30166241
- [Background] Dang UJ, Ziemba M, Clemens PR, Hathout Y, Conklin LS; CINRG Vamorolone 002/003 Investigators; Hoffman EP. Serum biomarkers associated with baseline clinical severity in young steroid-naive Duchenne muscular dystrophy boys. Hum Mol Genet. 2020 Aug 29;29(15):2481-2495. doi: 10.1093/hmg/ddaa132. PMID 32592467
- [Background] Ziemba M, Barkhouse M, Uaesoontrachoon K, Giri M, Hathout Y, Dang UJ, Gordish-Dressman H, Nagaraju K, Hoffman EP. Biomarker-focused multi-drug combination therapy and repurposing trial in mdx mice. PLoS One. 2021 Feb 22;16(2):e0246507. doi: 10.1371/journal.pone.0246507. eCollection 2021. PMID 33617542
- [Background] Dadgar S, Wang Z, Johnston H, Kesari A, Nagaraju K, Chen YW, Hill DA, Partridge TA, Giri M, Freishtat RJ, Nazarian J, Xuan J, Wang Y, Hoffman EP. Asynchronous remodeling is a driver of failed regeneration in Duchenne muscular dystrophy. J Cell Biol. 2014 Oct 13;207(1):139-58. doi: 10.1083/jcb.201402079. PMID 25313409
- [Background] Heier CR, Damsker JM, Yu Q, Dillingham BC, Huynh T, Van der Meulen JH, Sali A, Miller BK, Phadke A, Scheffer L, Quinn J, Tatem K, Jordan S, Dadgar S, Rodriguez OC, Albanese C, Calhoun M, Gordish-Dressman H, Jaiswal JK, Connor EM, McCall JM, Hoffman EP, Reeves EK, Nagaraju K. VBP15, a novel anti-inflammatory and membrane-stabilizer, improves muscular dystrophy without side effects. EMBO Mol Med. 2013 Oct;5(10):1569-85. doi: 10.1002/emmm.201302621. Epub 2013 Sep 9. PMID 24014378
- [Background] Damsker JM, Dillingham BC, Rose MC, Balsley MA, Heier CR, Watson AM, Stemmy EJ, Jurjus RA, Huynh T, Tatem K, Uaesoontrachoon K, Berry DM, Benton AS, Freishtat RJ, Hoffman EP, McCall JM, Gordish-Dressman H, Constant SL, Reeves EK, Nagaraju K. VBP15, a glucocorticoid analogue, is effective at reducing allergic lung inflammation in mice. PLoS One. 2013 May 7;8(5):e63871. doi: 10.1371/journal.pone.0063871. Print 2013. PMID 23667681
- [Background] Freishtat RJ, Nino G, Tsegaye Y, Alcala SE, Benton AS, Watson AM, Reeves EK, Haider SK, Damsker JM. Pharmacologically-induced mitotic synchrony in airway epithelial cells as a mechanism of action of anti-inflammatory drugs. Respir Res. 2015 Oct 29;16:132. doi: 10.1186/s12931-015-0293-4. PMID 26511361
- [Background] Dillingham BC, Knoblach SM, Many GM, Harmon BT, Mullen AM, Heier CR, Bello L, McCall JM, Hoffman EP, Connor EM, Nagaraju K, Reeves EKM, Damsker JM. VBP15, a novel anti-inflammatory, is effective at reducing the severity of murine experimental autoimmune encephalomyelitis. Cell Mol Neurobiol. 2015 Apr;35(3):377-387. doi: 10.1007/s10571-014-0133-y. Epub 2014 Nov 13. PMID 25392236
- [Background] Garvin LM, Chen Y, Damsker JM, Rose MC. A novel dissociative steroid VBP15 reduces MUC5AC gene expression in airway epithelial cells but lacks the GRE mediated transcriptional properties of dexamethasone. Pulm Pharmacol Ther. 2016 Jun;38:17-26. doi: 10.1016/j.pupt.2016.04.004. Epub 2016 Apr 29. PMID 27133900
- [Background] Damsker JM, Conklin LS, Sadri S, Dillingham BC, Panchapakesan K, Heier CR, McCall JM, Sandler AD. VBP15, a novel dissociative steroid compound, reduces NFkappaB-induced expression of inflammatory cytokines in vitro and symptoms of murine trinitrobenzene sulfonic acid-induced colitis. Inflamm Res. 2016 Sep;65(9):737-43. doi: 10.1007/s00011-016-0956-8. Epub 2016 Jun 3. PMID 27261270

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Started | 10 | 10 | 6 | 6 | 6 | 16
Completed | 10 | 10 | 6 | 6 | 6 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6 | Total
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 6 | 6 | 6 | 16 | 54
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 10 | 10 | 6 | 6 | 6 | 16 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 10 | 10 | 6 | 3 | 4 | 14 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 1 | 1 | 2 | 2 | 3 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White | 5 | 8 | 5 | 3 | 3 | 13 | 37
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 10 | 6 | 6 | 6 | 16 | 54
Age at first symptom [Mean (Standard Deviation); unit: months] | 20.8 (5.67) | 14.2 (4.47) | 30.0 (15.18) | 51.0 (23.92) | 32.2 (14.26) | 42.8 (27.59) | 31.7 (21.88)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events as Assessed by Common Terminology Criteria for Adverse Events Version 4.03 (CTCAE v4.03)
Description: An Adverse Event is any untoward medical occurrence in a subject and does not necessarily have to have a causal relationship with the intervention. Pre-existing conditions that worsen during the study are to be reported as AEs.
Time Frame: From the date of the subject's written informed consent until the final Week 16 Visit or the subject's participation in the study was completed
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
Participants | 7 | 9 | 6 | 4 | 3 | 12

2. Primary Outcome: Number of Participants With Drug Related Adverse Events as Assessed by Common Terminology Criteria for Adverse Events Version 4.03 (CTCAE v4.03)
Description: Drug related Adverse Events are TEAEs whose Causality were labeled as 'DEFINITE', 'POSSIBLE' or 'PROBABLE
Time Frame: as for outcome 1
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
Participants | 1 | 7 | 3 | 4 | 1 | 8

3. Primary Outcome: Number of Participants With Severe Adverse Events as Assessed by Common Terminology Criteria for Adverse Events Version 4.03 (CTCAE v4.03)
Description: Severe or medically significant but not immediately life -threatening: hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living; incapacitating with inability to work or perform normal daily activity.
Time Frame: as for outcome 1
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
Participants | 0 | 0 | 0 | 1 | 0 | 1

4. Primary Outcome: Number of Participants With Serious Adverse Events as Assessed by Common Terminology Criteria for Adverse Events Version 4.03 (CTCAE v4.03)
Description: A Serious Adverse Event (SAE) is defined as any AE regardless of causality that meets any of the following criteria:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of an existing hospitalization
  * Results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions
  * Results in a congenital anomaly/birth defect
  * Is an important medical event that may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above
Time Frame: From the date of the subject's written informed consent until the final Week 16 Visit or the subject's participation in the study was completed (SAEs through 30 days after final dose of study drug)
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
Participants | 0 | 0 | 0 | 1 | 0 | 1

5. Primary Outcome: Number of Participants With Adverse Events as Assessed by Common Terminology Criteria for Adverse Events Version 4.03 (CTCAE v4.03) Leading to Study Treatment Discontinuation
Description: Adverse Events leading to Study treatment discontinuation
Time Frame: as for outcome 1
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
Participants | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Change in Height (Absolute) From Baseline to Week 12
Description: Standing height will be assessed for subjects ages 2-<4 years; height calculated from ulnar length in subjects ages 7-<18.
Time Frame: Baseline, 12 weeks
Population: Safety set
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
cm | 1.98 (1.146) | 2.35 (0.568) | 0.55 (0.557) | 2.29 (1.609) | 0.60 (0.594) | 1.27 (1.313)

7. Primary Outcome: Change in Height (Percentile) From Baseline to Week 12
Description: as for outcome 6
Time Frame: Baseline, 12 weeks
Population: Safety set
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
percentile | 1.17 (11.538) | 2.09 (5.634) | -3.89 (3.907) | 2.02 (8.338) | -3.69 (3.408) | -0.30 (1.390)

8. Primary Outcome: Change in Height (Z-score) From Baseline to Week 12
Description: Standing height will be assessed for subjects ages 2-<4 years; height calculated from ulnar length in subjects ages 7-<18. The z-score (standard score) is the number of standard deviations by which the outcome measure is above or below the value in the general population. A Z-score of 0 represents the population mean. A measure above the normal value has a positive z-score (higher height).
Time Frame: Baseline, 12 weeks
Population: Safety set
Measure: Mean (Standard Deviation); unit: Z-score (score on a scale)
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
Z-score (score on a scale) | 0.04 (0.361) | 0.14 (0.201) | -0.12 (0.111) | 0.07 (0.253) | -0.13 (0.159) | 0.00 (0.194)

9. Primary Outcome: Change in Weight (Absolute) From Baseline to Week 12
Description: Body weight will be assessed at each of the scheduled time points.
Time Frame: Baseline, 12 weeks
Population: Safety set
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
kg | 0.43 (0.776) | 0.65 (0.911) | -0.18 (3.259) | 3.47 (3.133) | 1.53 (1.188) | 1.94 (2.598)

10. Primary Outcome: Change in Weight (Percentile) From Baseline to Week 12
Description: Body weight will be assessed at each of the scheduled time points.
Time Frame: Baseline, 12 weeks
Population: Safety set
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
percentile | -1.44 (12.835) | -1.97 (12.504) | -4.00 (11.672) | 15.20 (2.083) | 2.12 (4.235) | 4.22 (8.566)

11. Primary Outcome: Change in Weight (Z-score) From Baseline to Week 12
Description: Body weight will be assessed at each of the scheduled time points. The z-score (standard score) is the number of standard deviations by which the outcome measure is above or below the value in the general population. A Z-score of 0 represents the population mean. A measure above the normal value has a positive z-score (higher weight).
Time Frame: Baseline, 12 weeks
Population: Safety set
Measure: Mean (Standard Deviation); unit: Z-score (score on a scale)
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
Z-score (score on a scale) | -0.01 (0.406) | 0.05 (0.430) | -0.03 (0.438) | 0.55 (0.159) | 0.11 (0.147) | 0.22 (0.353)

12. Primary Outcome: Change in Body Mass Index (BMI) (Absolute) From Baseline to Week 12
Description: Body Mass Index is a measure of weight adjusted for height.
Time Frame: Baseline, Week 12
Population: Safety set
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
kg/m2 | -0.09 (0.933) | -0.04 (0.665) | 0.05 (1.394) | 1.53 (1.385) | 0.82 (0.784) | 0.60 (1.471)

13. Primary Outcome: Change in Body Mass Index (BMI) (Percentile) From Baseline to Week 12
Description: Body Mass Index is a measure of weight adjusted for height.
Time Frame: Baseline, Week 12
Population: Safety set
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
percentile | -2.85 (24.623) | -1.61 (12.509) | -3.00 (15.781) | 10.78 (7.312) | 6.22 (6.849) | 4.44 (11.498)

14. Primary Outcome: Change in Body Mass Index (BMI) (Z-score) From Baseline to Week 12
Description: Body Mass Index is a measure of weight adjusted for height. The z-score (standard score) is the number of standard deviations by which the outcome measure is above or below the value in the general population. A Z-score of 0 represents the population mean. A measure above the normal value has a positive z-score (higher BMI).
Time Frame: Baseline, Week 12
Population: Safety set
Measure: Mean (Standard Deviation); unit: Z-score (score on a scale)
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
Z-score (score on a scale) | -0.05 (0.764) | -0.02 (0.495) | 0.27 (0.771) | 1.10 (0.584) | 0.29 (0.317) | 0.29 (0.483)

15. Primary Outcome: Change in Diastolic Blood Pressure
Description: Change from Baseline to Week 12 in diastolic sitting blood pressure.
Time Frame: Day 1, Week 2, Week 6, Week 12, Week 16
Population: Safety set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
mmHg | -0.44 (8.248) | 2.00 (8.179) | -3.17 (7.333) | 5.80 (6.979) | 1.50 (6.950) | -2.40 (11.915)

16. Primary Outcome: Change in Systolic Blood Pressure
Description: Change from Baseline to Week 12 in systolic sitting blood pressure.
Time Frame: Day 1, Week 2, Week 6, Week 12, Week 16
Population: Safety set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
mmHg | -2.33 (12.923) | -2.20 (11.233) | -2.50 (6.504) | 5.00 (13.266) | 2.50 (5.958) | 0.07 (11.591)

17. Primary Outcome: Number of Participants With Treatment Emergent Cushingoid Features
Description: Treatment emergent cushingoid features based on physical examination at all baseline, on-treatment and post-treatment assessments
Time Frame: Baseline through Week 16
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
Participants | 0 | 0 | 0 | 1 | 0 | 0

18. Primary Outcome: Number of Participants With Clinically Significant Treatment-emergent Abnormal Clinical Laboratory Test Result
Description: Each subject had blood drawn and urine collected for the standard hematology, chemistry and lipids clinical laboratory tests. In addition, fasting glucose and insulin, morning cortisol, as well as, in the additional 12 to <18 years age group, LH, FSH, TSH, FT4 were collected. HbA1c determination had also to be performed if urine glucose was positive and/or fasted glucose levels was above normal limits. Any treatment-emergent clinically significant abnormal laboratory test result was reporte
Time Frame: Day 1, Week 6, Week 12, Week 16
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
Participants
  Cortisol decreased | 0 | 1 | 2 | 0 | 0 | 2
  Blood glucose decreased | 0 | 0 | 0 | 0 | 0 | 1
  Blood insulin increased | 0 | 0 | 0 | 0 | 0 | 1
  Blood TSH increased | 0 | 0 | 0 | 0 | 0 | 1
  Tyroxin free increased | 0 | 0 | 0 | 0 | 0 | 1

19. Primary Outcome: Categorical Analysis of QTcF at Week 12
Description: 12-lead 1electrocardiogram (ECG) as recorded after subject has rested quietly in a supine position for at least 5 minutes. ECG components are QRS duration, PR [PQ] interval, RR interval, QT interval and QTc.
Time Frame: Baseline, Week 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 5 | 15
Participants
  =< 450 msec | 10 | 10 | 6 | 6 | 5 | 15
  > 450 msec | 0 | 0 | 0 | 0 | 0 | 0

20. Primary Outcome: Number of Eyes With Cataract
Description: Cataract was diagnosed by the presence of partial or complete opacity of the crystalline lens at Baseline and Week 12.
Time Frame: Baseline - Week 12
Population: Safety set
Measure: Number; unit: eyes
Units Other Than Participants: eye
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 9 | 10 | 6 | 6 | 6 | 16
Number analyzed (eye) | 18 | 19 | 12 | 12 | 12 | 32
eyes
  No Cataract : Baseline | 18 | 19 | 12 | 12 | 8 | 17
  No Cataract : Week 12: number analyzed (Participants) | 9 | 4 | 6 | 5 | 5 | 14
  No Cataract : Week 12: number analyzed (eye) | 18 | 8 | 12 | 10 | 10 | 28
  No Cataract : Week 12 | 18 | 8 | 12 | 10 | 8 | 15
  Cataract : Baseline | 0 | 0 | 0 | 0 | 4 | 15
  Cataract : Week 12: number analyzed (Participants) | 9 | 4 | 6 | 5 | 5 | 14
  Cataract : Week 12: number analyzed (eye) | 18 | 8 | 12 | 10 | 10 | 28
  Cataract : Week 12 | 0 | 0 | 0 | 0 | 2 | 13

21. Primary Outcome: Number of Eyes With Glaucoma
Description: Glaucoma was diagnosed by ocular pressure at Baseline and Week 12.
Time Frame: Baseline - Week 12
Population: Safety set
Measure: Number; unit: eyes
Units Other Than Participants: eye
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 9 | 10 | 6 | 6 | 6 | 16
Number analyzed (eye) | 18 | 19 | 12 | 12 | 12 | 32
eyes
  No Glaucoma: Baseline: number analyzed (Participants) | 9 | 10 | 6 | 6 | 4 | 10
  No Glaucoma: Baseline: number analyzed (eye) | 18 | 19 | 12 | 12 | 8 | 19
  No Glaucoma: Baseline | 18 | 19 | 12 | 12 | 8 | 17
  No Glaucoma: Week 12: number analyzed (Participants) | 9 | 4 | 6 | 5 | 4 | 8
  No Glaucoma: Week 12: number analyzed (eye) | 18 | 8 | 12 | 10 | 8 | 15
  No Glaucoma: Week 12 | 18 | 8 | 12 | 10 | 8 | 15
  Suspected Glaucoma: Baseline: number analyzed (Participants) | 9 | 10 | 6 | 6 | 4 | 10
  Suspected Glaucoma: Baseline: number analyzed (eye) | 18 | 19 | 12 | 12 | 8 | 19
  Suspected Glaucoma: Baseline | 0 | 0 | 0 | 0 | 0 | 2
  Suspected Glaucoma: Week 12: number analyzed (Participants) | 9 | 4 | 6 | 5 | 4 | 8
  Suspected Glaucoma: Week 12: number analyzed (eye) | 18 | 8 | 12 | 10 | 8 | 15
  Suspected Glaucoma: Week 12 | 0 | 0 | 0 | 0 | 0 | 0
  Glaucoma: Baseline: number analyzed (Participants) | 9 | 10 | 6 | 6 | 4 | 10
  Glaucoma: Baseline: number analyzed (eye) | 18 | 19 | 12 | 12 | 8 | 19
  Glaucoma: Baseline | 0 | 0 | 0 | 0 | 0 | 0
  Glaucoma: Week 12: number analyzed (Participants) | 9 | 4 | 6 | 5 | 4 | 8
  Glaucoma: Week 12: number analyzed (eye) | 18 | 8 | 12 | 10 | 8 | 15
  Glaucoma: Week 12 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Pre-dose and Post-dose Plasma Concentration Measurements of Vamorolone at Day 1 and Week 2
Description: The plasma concentration of vamorolone was measured on Day 1 and Week 2 predose, and 1h, 2h and 6h postdose and also 4h and 8h post in the 7-18 year groups.
Time Frame: Day 1, Week 2
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng / mL
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
ng / mL
  Day 1 - predose | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Day 1 - 1h | 198.3 (196.67) | 471.3 (333.61) | 142.5 (225.74) | 519.1 (437.26) | 142.5 (225.74) | 519.1 (437.26)
  Day 1 - 2h | 236.7 (153.58) | 769.3 (527.67) | 216.4 (181.19) | 780.5 (457.91) | 216.4 (181.19) | 780.5 (457.91)
  Day 1 - 4h: number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 16
  Day 1 - 4h |  |  | 163.8 (103.74) | 711.1 (353.60) | 163.8 (103.74) | 711.1 (353.60)
  Day 1 - 6h | 125.7 (84.83) | 280.0 (249.99) | 148.0 (109.33) | 389.1 (307.57) | 148.0 (109.33) | 389.1 (307.57)
  Day 1 - 8h: number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 16
  Day 1 - 8h |  |  | 78.5 (41.66) | 170.6 (183.67) | 78.5 (41.66) | 170.6 (183.67)
  Week 2 - predose | 0.0 (0.00) | 0.0 (0.00) | 0.7 (2.06) | 2.9 (5.22) | 0.7 (2.06) | 2.9 (5.22)
  Week 2 - 1h | 346.0 (329.08) | 409.8 (385.65) | 192.0 (199.92) | 463.7 (348.19) | 192.0 (199.92) | 463.7 (348.19)
  Week 2 - 2h | 360.4 (222.93) | 829.4 (740.83) | 217.8 (149.31) | 686.3 (369.69) | 217.8 (149.31) | 686.3 (369.69)
  Week 2 - 4h: number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 16
  Week 2 - 4h |  |  | 207.6 (167.99) | 603.0 (346.88) | 207.6 (167.99) | 603.0 (346.88)
  Week 2 - 6h | 134.5 (110.99) | 272.0 (109.71) | 158.9 (105.34) | 300.2 (206.18) | 158.9 (105.34) | 300.2 (206.18)
  Week 2 - 8h: number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 16
  Week 2 - 8h |  |  | 55.8 (31.81) | 174.7 (137.78) | 55.8 (31.81) | 174.7 (137.78)

23. Secondary Outcome: Descriptive Statistics of PK Parameters - Tmax
Description: Tmax is the time to reach the maximum observed concentration collected during a dosing interval
Time Frame: Day 1, Week 2
Population: PK analysis set
Measure: Median (Full Range); unit: h
Groups:
- Group 1: Patients aged 2-<4 years receiving oral Vamorolone at 2.0 mg/kg/day for 12 weeks.
- Group 2: Patients aged 2-<4 years receiving oral Vamorolone at 6.0 mg/kg/day for 12 weeks.
- Group 3: Patients aged 7-<18 years receiving oral Vamorolone at 2.0 mg/kg/day for 12 weeks.
- Group 4: Patients aged 7-<18 years receiving oral Vamorolone at 6.0 mg/kg/day for 12 weeks.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 10 | 10 | 12 | 22
h
  Day 1 | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 6.0]
  Week 2: number analyzed (Participants) | 9 | 8 | 12 | 22
  Week 2 | 1.9 [1.0 to 6.3] | 2.0 [1.1 to 6.0] | 2.9 [1.0 to 8.0] | 2.0 [1.0 to 6.0]

24. Secondary Outcome: Descriptive Statistics of PK Parameters - Cmax
Description: Cmax is the maximum observed concentration
Time Frame: Day 1, Week 2
Population: PK analysis set
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 10 | 10 | 12 | 22
ng/mL
  Day 1 | 246.8 (2.01) | 781.7 (1.77) | 254.5 (2.04) | 922.2 (1.60)
  Week 2: number analyzed (Participants) | 9 | 8 | 12 | 22
  Week 2 | 349.3 (2.06) | 719.5 (2.23) | 334.5 (1.67) | 765.5 (1.59)

25. Secondary Outcome: Descriptive Statistics of PK Parameters in Subjects Aged 2 to 4 Years - AUC 0-6
Description: AUC 0-6 is the area under the concentration-time curve during the first 6 hours after dosing
Time Frame: Day 1, Week 2
Population: PK analysis set - Subjects aged 2 to 4 years
Measure: Geometric Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 8 | 8
ng.h/mL
  Day 1 | 816.3 (1.72) | 2216.2 (1.47)
  Week 2: number analyzed (Participants) | 7 | 7
  Week 2 | 1448.4 (1.38) | 2571.6 (2.02)

26. Secondary Outcome: Descriptive Statistics of PK Parameters in Subjects Aged 7 to 18 Years - AUC 0-inf
Description: AUC 0-8 is the area under the concentration-time curve after dosing extrapolated to infinity
Time Frame: Day 1, Week 2
Population: PK analysis set - subjects aged 7 to 18 years
Measure: Geometric Mean (Standard Deviation); unit: ng.h/mL
Groups:
- Group 3: Patients aged 7-<18 years receiving oral Vamorolone at 2.0 mg/kg/day for 12 weeks. This Group is combining subjects from Treatment groups 3 and 5.
- Group 4: Patients aged 7-<18 years receiving oral Vamorolone at 6.0 mg/kg/day for 12 weeks. This Group is combining subjects from Treatment groups 4 and 6.
Arm/Group | Group 3 | Group 4
Number analyzed (Participants) | 6 | 13
ng.h/mL
  Day 1: number analyzed (Participants) | 5 | 13
  Day 1 | 1253.0 (1.65) | 4119.8 (1.53)
  Week 2: number analyzed (Participants) | 6 | 9
  Week 2 | 1528.6 (1.15) | 3587.7 (1.72)

27. Other Pre Specified Outcome: Change From Baseline to Week 12 in Bayley-III Gross Motor Scale (Ages 2 to <4 Years Only)
Description: The Bayley-III Gross Motor scale is a functional assessment, an accurate reflection of muscle strength for subjects with DMD ages 2 to <4 years. The minimum score value is 0 and the maximum score value is 72. Higher scores mean a better outcome.
Time Frame: Baseline, Week 12
Population: Safety set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group 1 | Treatment Group 2
Number analyzed (Participants) | 9 | 10
score on a scale | 0.44 (1.130) | 2.50 (1.716)

28. Other Pre Specified Outcome: Change From Baseline to Week 12 in Morning Cortisol Concentration
Description: Morning cortisol [adrenal suppression] samples were collected after the subject has fasted for ≥ 6 hours and prior to administration of the daily dose of study medication at Day 1 and Week 12 Visits, before 10 AM local time
Time Frame: Baseline, Week 12
Population: Safety set
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 8 | 6 | 6 | 6 | 15
nmol/L | -184.700 (138.2020) | -217.750 (103.9832) | -110.667 (85.8596) | -248.667 (186.9060) | 12.000 (49.3356) | -34.933 (42.1485)

29. Other Pre Specified Outcome: Change From Baseline to Week 12 in Bone Turnover Biomarkers (Serum Type 1 Collagen C-telopeptide [CTX1])
Description: Samples for CTX1, osteocalcin and P1NP were collected at the Day 1 and Week 12 Visits after the subject has fasted for ≥ 6 hours and prior to administration of the daily dose of study medication
Time Frame: Baseline, Week 12
Population: Safety set
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 9 | 6 | 5 | 6 | 13
ng/L | 28.300 (387.1423) | 138.000 (257.6640) | 93.500 (235.7446) | 101.800 (365.3542) | 631.833 (155.3621) | 273.000 (335.4937)

30. Other Pre Specified Outcome: Change From Baseline to Week 12 in Bone Turnover Biomarkers (Osteocalcin)
Description: as for outcome 29
Time Frame: Baseline, Week 12
Population: Safety set
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 9 | 6 | 5 | 6 | 13
ug/L | -3.340 (21.0550) | 2.422 (10.6960) | 14.817 (18.7328) | -1.120 (15.8528) | 31.700 (11.6915) | 16.546 (9.1486)

31. Other Pre Specified Outcome: Change From Baseline to Week 12 in Bone Turnover Biomarkers (Serum Aminoterminal Propeptide of Type I Collagen [P1NP] )
Description: as for outcome 29
Time Frame: Baseline, Week 12
Population: Safety set
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 9 | 6 | 5 | 6 | 14
ug/L | -39.870 (188.7787) | 14.478 (117.5704) | 19.067 (78.6139) | -82.840 (178.0726) | 318.850 (99.0038) | 149.671 (106.2874)

32. Other Pre Specified Outcome: Change From Baseline to Week 12 in Insulin Resistance Biomarkers (Glucose)
Description: Glucose, HbA1c and insulin were collected at the Day 1 and Week 12 Visits after the subject has fasted for ≥ 6 hours and prior to administration of the daily dose of study medication.
Time Frame: Baseline, Week 12
Population: Safety set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 16
mmol/L | -0.160 (0.2912) | -0.243 (0.6309) | -0.063 (0.3524) | -0.335 (0.3815) | 0.195 (0.5727) | -0.254 (0.3909)

33. Other Pre Specified Outcome: Change From Baseline to Week 12 in Insulin Resistance Biomarkers (Hemoglobin A1c [HbA1c])
Description: Glucose, HbA1c and insulin were collected at the Day 1 and Week 12 Visits after the subject has fasted for ≥ 6 hours and prior to administration of the daily dose of study medication. The Baseline sample for HbA1c measurement may have been collected non-fasting.
Time Frame: Baseline, Week 12
Population: Safety set
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Number analyzed (Participants) | 9 | 9 | 5 | 6 | 5 | 11
percent | 0.1 (0.26) | 0.0 (0.15) | 0.0 (0.16) | 0.0 (0.10) | 0.0 (0.11) | -0.1 (0.12)

34. Other Pre Specified Outcome: Change From Baseline to Week 12 in Insulin Resistance Biomarkers (Insulin)
Description: as for outcome 32
Time Frame: Baseline, Week 12
Population: Safety set - No subjects were analyzed in Group 1 and 5
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 6
Number analyzed (Participants) | 9 | 3 | 6 | 9
pmol/L | 6.333 (20.5183) | 0.667 (33.0051) | 46.333 (51.9256) | -26.333 (51.1493)

ADVERSE EVENTS:
Time Frame: AEs were collected through Week 16 Visit or the subject's participation in the study was completed (SAEs through 30 days after final dose study drug).
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/6 | 0/6 | 0/6 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/6 | 1/6 | 0/6 | 1/16
Other Adverse Events (participants affected / at risk) | 7/10 | 9/10 | 6/6 | 4/6 | 3/6 | 11/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group 1 (N=10) | Treatment Group 2 (N=10) | Treatment Group 3 (N=6) | Treatment Group 4 (N=6) | Treatment Group 5 (N=6) | Treatment Group 6 (N=16)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group 1 (N=10) | Treatment Group 2 (N=10) | Treatment Group 3 (N=6) | Treatment Group 4 (N=6) | Treatment Group 5 (N=6) | Treatment Group 6 (N=16)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal suppression (Endocrine disorders) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Energy increased (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (8) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood insulin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cortisol decreased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Thyroxine free increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 4 (5)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Behaviour disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Compulsive lip biting (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disruptive mood dysregulation disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT05185622/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT05185622/SAP_001.pdf